CLINICAL TRIAL: NCT02689778
Title: Effect of Pirfenidone on Glomerular Filtration Rate and Albuminuria in Patients With Diabetic Nephropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Grupo Medifarma, S. A. de C. V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1497
Record Dates: First submitted 2016-02-12; First posted 2016-02-24 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2019-08

CONDITIONS: Diabetic Nephropathy; Albuminuria
Keywords: Pirfenidone; Diabetic nephropathy
MeSH Terms: conditions — Diabetic Nephropathies; Albuminuria | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pirfenidone (Experimental): Oral pirfenidone 600 mg with breakfast and 1200 mg with dinner for 12 months.
  Interventions: Drug: Pirfenidone
- Placebo (Placebo Comparator): Oral placebo with breakfast and with dinner for 12 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Oral pirfenidone 600 mg with breakfast and 1200 mg pirfenidone with dinner for 12 months.
  Other Names: Kitoscell LP
  Arms: Pirfenidone
Drug: Placebo — Identical tablets without active substance
  Arms: Placebo

SUMMARY:
It is estimated that approximately 30% of patients with diabetes develop diabetic nephropathy. Diabetic nephropathy is a multifactorial progressive disease that occurs through various mechanisms such as hyperglycemia, oxidative stress, inflammation and fibrosis, control or blocking these mechanisms are therefore potential therapeutical targets for this entity. Current treatment options are based on the glycemic control, blood pressure control, as well as the use of medications such as angiotensin-converting enzyme inhibitors and Angiotensin II receptor antagonists, these actions are not enough to stop progression. Pirfenidone is a drug with antifibrotic, antioxidant, and anti-inflammatory properties. Although the specific mechanism is unknown, pirfenidone interferes with the expression, secretion and the effect of the β (TGF-β) transforming growth factor. The investigators plan to carry out a controlled clinical study to evaluate the effect of pirfenidone in patients with type 2 diabetes and nephropathy. The period of time the treatment will be administered will be of 12 months, 62 patients will be included. The primary outcome will be improvement in glomerular filtration rate. The secondary outcomes will be number of patients requiring replacement therapy, 24 hour urine microalbuminuria and change in the concentration of TGF - β. Change in these parameters will be evaluated at the end of the treatment period (12 months). Throughout the study the incidence of adverse events will be recorded, wich will allow us to learn about the safety and security of the drug in this population.

ELIGIBILITY:
Inclusion criteria

* Body mass index (BMI) less than 35 kg/m2
* Diagnosis of diabetes mellitus type 2
* Glomerular filtration rate of 15-89 ml/min
* Albuminuria ≥30 mg/24 h and < 3.5 g/24 h
* Individuals with blood pressure less than 140/90 mmHg or treated with stable doses of anti-hypertensive drugs.
* Glycated hemoglobin <10%

Exclusion criteria

* Another etiology of renal disease (autoimmune diseases, polycystic kidney disease)
* Repeated urinary tract infections (more than three episodes in the past year)
* Photosensitivity to any drug
* Liver disease
* Pregnancy
* Breastfeeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-03; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Effect of oral pirfenidone (1800 mg) in albuminuria | 12 months
Effect of oral pirfenidone (1800 mg) in glomerular filtration rate | 12 months

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | 12 months
  hypersensitivity, photosensitivity, liver function test alteration

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (INCMNSZ), Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No